CLINICAL TRIAL: NCT02198521
Title: Staged Bilateral Carpal Tunnel Release: Which Side Hurts More?
Status: Withdrawn | Type: Observational
Why Stopped: The researcher and principal investigator working on this study left the institution.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, MD/PhD, Massachusetts General Hospital
Other Study IDs: 2009P001019 AME 339
Record Dates: First submitted 2014-06-10; First posted 2014-07-23 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Carpal Tunnel Syndrome; Pain
Keywords: Patients undergoing staged bilateral open Carpal Tunnel Release (CTR) have no difference in overall pain intensity of pain between sides.
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bilateral Carpal Tunnel Syndrome (CTS)

SUMMARY:
Title Staged Bilateral Carpal Tunnel Release: Which Side Hurts More? Primary null hypothesis Patients undergoing staged bilateral open Carpal Tunnel Release (CTR) have no difference in overall pain intensity of pain between sides.

Secondary null hypotheses

* There is no correlation in overall pain intensity after open CTR surgery and distal sensory latency, distal motor latency, electromyography (EMG), demographics, occupation, avocation, relevant comorbidities, dominance, left vs. right, Pain Self-Efficacy, Patient Reported Outcomes Measurement Information System (PROMIS) Upper Extremity or PROMIS depression when both surgeries are performed within 6 months.
* There is no difference in satisfaction with treatment at the time of suture removal after the first and second open CTR surgery when both are performed within 6 months..

IRB: 2009-p-001-019 ClinicalTrials.gov: Not mandatory, (b/o observational) Authors: Drijkoningen, Braun, Ring Journal: To be discussed Design: Prospective cohort study Background Many hand surgeons note that patients undergoing staged bilateral open carpal tunnel release often experience more pain with the second side. The investigator felt this was an easily testable hypothesis worthy of study.

Subjects

Eligibility:

Inclusion:

* Age 18 or older
* Idiopathic carpal tunnel syndrome
* No prior surgery for carpal tunnel syndrome

Exclude:

* Pregnant women
* Not fluent in English

Response Variables:

* 11-point ordinal measure of overall pain intensity during and after surgery measured at the time of suture removal.
* 11-point ordinal measure of satisfaction with treatment
* PROMIS upper extremity

Explanatory Variables:

* Distal Sensory Latency (DSL)
* Distal Motor Latency (DML)
* EMG changes
* Demographics: age, sex, race, occupation, avocation
* Time limit between two surgeries < 6 months
* Relevant comorbidities: Trapeziometacarpal (TMC) arthrosis, ulnar neuropathy, trigger finger
* Involved hand (Dominance, Side)
* First side vs. second side surgery
* PROMIS Pain Interference Computer Adaptive Testing (CAT)
* Pain Self Efficacy Questionnaire (PSEQ-2)
* PROMIS Depression

Methods The investigator and study staff will invite all adult patients (age 18 and older) presenting to the Orthopaedic Hand and Upper Extremity Service Department at Massachusetts General Hospital (MGH) with bilateral carpal tunnel syndrome planning staged bilateral carpal tunnel release.

Analysis Power analysis An a priori power analysis for matched pairs was performed. To detect the difference between two dependent means an effect size of 0.5 at alpha of 0.05 and 80% power, a total sample size of 34 patients is needed.As the investigator expects to have patients who will be lost to follow-up the investigators will count 10% extra, a total of 38 patients will be needed.

Univariate analysis: Variables will be presented with frequencies and percentages for categorical variables and as mean with standard deviation or median with interquartile range for respectively normal or non-normal distributed continuous variables. Normality of continuous distributed variables will be tested a paired T-Test.

Bivariate and multivariable analysis will be performed and subsequently all variables with a probability < 0.10 in bivariate analysis will be inserted in a backward, stepwise, multivariable linear regression analysis to assess their ability to explain variation in outcome. The 11 point Likert Pain scale score is considered significant when there is a difference of more than 1.4 points (2.8 SD*0.5 effect size)on a scale from 1-10.[9]

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Idiopathic carpal tunnel syndrome
* No prior surgery for carpal tunnel syndrome

Exclusion Criteria:

* Pregnant women
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bilateral CTS patients undergoing bilateral carpal tunnel release
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09

PRIMARY OUTCOMES:
Overall Pain Intensity | 2 weeks after surgery within 6 month timeframe
  The overall pain intensity is measured on an 11-point ordinal measure of overall pain intensity after surgery measured at the time of suture removal.

SECONDARY OUTCOMES:
Overall Satisfaction | 2 weeks after surgery within a 6 month timeframe
  11-point ordinal measure of satisfaction with treatment measured 2 weeks after surgery during suture removal
Patient Reported Outcome for Upper Extremity Function | 2 weeks after surgery within 6 month timeframe
  PROMIS upper extremity
Electromyogram Results | Before Surgery
  EMG DSL and DML
Demographics | 2 weeks after first surgery
  Age, sex, race, occupation, avocation
Comorbidities | 2 weeks after surgery
  Relevant comorbidities: TMC Arthrosis, ulnar neuropathy, trigger finger
Hand Dominance and Side of Surgery | 2 weeks after surgery
Patient Reported Pain Interference | 2 weeks after surgery within 6 month timeframe
  PROMIS Pain Interference (CAT)
Patient Self Efficacy Questionnaire | 2 weeks after surgery within 6 month timeframe
  PSEQ-2
Patient Reported Depression | 2 weeks after surgery within 6 month timeframe
  PROMIS Depression

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States